CLINICAL TRIAL: NCT02248454
Title: Evaluation of Insulin Bolus for High Fat Meals
Brief Title: Insulin Bolus Required for High Fat Foods in Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Joslin Diabetes Center (Other)
Collaborators: Boston Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: High fat bolus
Record Dates: First submitted 2014-09-22; First posted 2014-09-25 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2017-04

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Lispro

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Insulin bolus dose/type (Experimental): Lispro insulin, dose calculated by modeling analysis
  Interventions: Drug: Lispro

INTERVENTIONS:
Drug: Lispro — Increasing insulin doses
  Other Names: Humalog

SUMMARY:
The purpose of this study is to evaluate an insulin bolus for use to cover higher fat meals.

Subjects will have several admissions during which the investigators will apply an iterative dose escalation protocol to derive an optimized insulin bolus dose (carbohydrate-to-insulin ratio for fat to minimize postprandial hyperglycemia following higher fat meals. The investigators hypothesize that the incremental insulin dose required to cover dietary fat in patients with type 1 diabetes will be related to total daily insulin dose (U/kg).

DETAILED DESCRIPTION:
Subjects for this study will be adults with type 1 diabetes who use an insulin pump for diabetes self-management.

Subjects will be admitted to the clinical research center in the morning in the fasting state. Subjects will have several admissions. During the initial two admissions, subjects will receive either pizza-low fat or pizza-high fat, covered with insulin doses calculated from their usual insulin-to-carbohydrate ratio. Study subjects in whom the bolus did not provide adequate insulin coverage for pizza-high fat will then undergo an additional 1-5 admissions during which they will receive the pizza-high fat meal with progressively increasing insulin doses until ≥ 90% of all postprandial glucose values are within the target range 80-180 mg/dL.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (aged 18-75 years) with type 1 diabetes > 3 years, on insulin pump therapy.

Exclusion Criteria:

* History or symptoms suggestive of gastroparesis or gastric dysmotility; History of celiac disease, pancreatic exocrine dysfunction or other conditions that cause malabsorption or maldigestion; Eating disorder; Diet allergies; Special diet restrictions, such as vegan; Medications know to affect insulin sensitivity (such as glucocorticoids) or affect gastrointestinal motility (such as reglan); High-titre insulin autoantibodies with delayed insulin kinetics; Women who are breast feeding, pregnant, or wanting to become pregnant.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-09; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Predictors of fat "sensitivity" | 0-360 minutes
  To test the hypothesis that incremental dose increase required to cover dietary fat in patients with type 1 diabetes will be related to total daily insulin dose (TDD; U/kg) we will perform regression analysis with TDD as independent variable and the increase in insulin requirements (calculated as percent change for high fat vs low fat meal) as the dependent variable.

CONTACTS AND LOCATIONS:
Overall Officials: Howard Wolpert, MD, Principal Investigator — Joslin Diabetes Center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bell KJ, Toschi E, Steil GM, Wolpert HA. Optimized Mealtime Insulin Dosing for Fat and Protein in Type 1 Diabetes: Application of a Model-Based Approach to Derive Insulin Doses for Open-Loop Diabetes Management. Diabetes Care. 2016 Sep;39(9):1631-4. doi: 10.2337/dc15-2855. Epub 2016 Jul 7. PMID 27388474